CLINICAL TRIAL: NCT03219086
Title: A Prospective Randomized Double Blind Comparison of 7,5 mg Hyperbaric Bupivacaine With 2,5mcg Sufentanyl or 50 mg Hyperbaric Prilocaine With 2,5 mcg Sufentanyl for Caesarean Sections
Brief Title: Spinal Prilocaine for Caesarian Sections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: AZ Klina (Other); AZ Middelheim (Unknown)
Responsible Party: Principal Investigator, Dr M. B. Breebaart, MD, PhD, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ec nr 17/07/77
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Combined Spinal Epidural Anesthesia; Prilocaine; Bupivacaine; Pain
Keywords: combined spinal epidural anesthesia; caesarian section; prilocaine; bupivacaine
MeSH Terms: conditions — Pain | interventions — Anesthesia, Spinal; Prilocaine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: prospective double blind randomised
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The spinal solution will be prepared by an independent anaesthetist, anaesthetist trainee or research nurse on a sterile table after opening the sealed envelope with the appointed study group. The patient, the anaesthetist performing the CSE and the observer are not aware of the local anaesthetic solution administered.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group M (Active Comparator): combined spinal epidural anesthesia with spinal administration of 7,5 mg hyperbaric bupivacaine 0,5% (Marcaine H) + 2,5mcg sufentanyl ( 5 mcg/ml)( Janssens -cilag) +1 ml nacl0,9%
  Interventions: Procedure: combined spinal epidural anaesthesia; Drug: Bupivacaine
- Group P (Active Comparator): A combined spinal epidural anesthesia with spinal administration of 50 mg hyperbaric prilocaine 2% (Tachipri, Nordic Pharma) + 2,5mcg sufentanyl (5 mcg/ml) (Janssens-cilag)
  Interventions: Procedure: combined spinal epidural anaesthesia; Drug: Prilocaine

INTERVENTIONS:
Procedure: combined spinal epidural anaesthesia — To give surgical anesthesia for performance of the caesarian section a combined spinal epidural anesthesia will be performed with different spinal solutions according to the appointed study group
  Other Names: CSE; Spinal anesthesia; prilocaine
Drug: Prilocaine — A combined spinal epidural anesthesia with spinal administration of 50 mg hyperbaric prilocaine 2% (Tachipri, Nordic Pharma) + 2,5mcg sufentanyl (5 mcg/ml) (Janssens-cilag)
  Other Names: Tachipri
  Arms: Group P
Drug: Bupivacaine — combined spinal epidural anesthesia with spinal administration of 7,5 mg hyperbaric bupivacaine 0,5% (Marcaine H) + 2,5mcg sufentanyl ( 5 mcg/ml)( Janssens -cilag) +1 ml nacl0,9%
  Other Names: Marcaine
  Arms: Group M

SUMMARY:
Prilocaine theoretically could provide faster onset because of its lower pKa (7,7) compared to bupivacaine (8,1). The primary objective of this prospective double blind randomized trial is to determine block onset of spinal hyperbaric prilocaine compared to bupivacaine, both with a small dose of sufentanyl as an additive.The primary hypothesis is that a significant larger amount of patients will gain surgical readiness within 8 minutes after spinal injection of prilocaine with sufentanyl compared to bupivacaine with sufentanyl. Surgical readiness is defined as a sensory block level of T5 tested by loss of cold sensation.

DETAILED DESCRIPTION:
This study is designed as a randomised prospective double blind multi centre study.

Following approval by the Hospital Ethics committee of the University Hospital Antwerp and all participating hospitals, all-in term (37-42 weeks of gestation) pregnant women planned for a caesarean section will be asked to participate in this trial.

Patients will be randomised to receive either spinal prilocaine with sufentanyl or spinal bupivacaine with sufentanyl.The patient, the anaesthetist performing the CSE and the observer are not aware of the local anaesthetic solution administered.

Preoperative a combined spinal epidural puncture will be performed in the sitting position at the level of L2-L3 or L3-L4 . Vital parameters will be registered at regular intervals. Block characteristics ( onset, duration and intensity of the sensory block and motor block) will be measured at regular intervals.

Patients with insufficient analgesia will receive a top up dose of 5 ml lidocaine 2 % via the epidural catheter.

Time of birth, neonatal outcome (Apgar score 1 min, 5 min and 10 minutes after birth) and admission to the nicu as well as umbilicus venous and arterial blood gasses are recorded.

Patients will be discharged from the PACU when motor block reached a Bromage score 1 Time intervals of discharge to the ward will be registered.At the maternity ward the time of first contact of the baby and the mother and first breast feed (if applicable) will be registered.

One week postoperative patients will be called and asked if they experienced any postoperative symptoms like headache, micturition problems or symptoms resembling Transient Neurological Symptoms

ELIGIBILITY:
Inclusion Criteria:

* A term Pregnant women (37-42 weeks)scheduled for caesarian section

Exclusion Criteria:

* Patient refusal
* Twin or multiple pregnancy
* Preeclampsia
* Contraindication neuraxial technique
* Indication general anaesthesia
* BMI before pregnancy >35
* Maternal height <155 cm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
onset time surgical readiness | from start spinal anaesthesia to start of surgery (up to 30 minutes)
  amount of minutes from spinal injection (T0) to loss of cold sensation on the fifth thoracic dermatome

SECONDARY OUTCOMES:
regression interval of the motor block | up to 3 hours
  Time from spinal injection to a Bromage score of 1 (knee flexion possible)
occurrence of hypotension | from spinal injection(T0) to motor block regression ( up to 3 hours)
  percentage of study group with hypotension defined as a systolic BP of less than 100 mm Hg or a 20% drop from the baseline level
sensory block level | Up to 3 hours
  highest dermatome measured during the study
discharge time maternity ward | Up to 3 hours
  the time interval from spinal injection (T0) to discharge to the maternity ward
First Breast feed | up to 6 hours
  the time interval from injection (T0) to first breast feeding

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - AZ Middelheim, Berchem, Antwerpen
  - AZ KLina, Brasschaat, Antwerp
  - University Hospital Antwerp, Antwerp